CLINICAL TRIAL: NCT05293860
Title: Effects of Connective Tissue Manipulation on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Hitit University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 499
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-06

CONDITIONS: Menopause Syndrome
Keywords: Menopause; Vasomotor symptom; Massage; Connective tissue massage; Connective tissue manipulation; Physiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Connective tissue manipulation (Experimental): Connective tissue manipulation will be applied to participants' back for 5-20 minutes, 3 times a week for 4 weeks in this group.
  Interventions: Other: Connective tissue manipulation
- Superficial massage with the head of the therapeutic ultrasound device (Sham Comparator): Superficial massage with the head of the therapeutic ultrasound device will be applied to participants' back for 15 minutes, 3 times a week for 4 weeks in this group.
  Interventions: Other: Superficial massage with the head of the therapeutic ultrasound device

INTERVENTIONS:
Other: Connective tissue manipulation — Connective tissue manipulation will be applied to participants' back for 5-20 minutes, 3 times a week for 4 weeks in this group.
  Arms: Connective tissue manipulation
Other: Superficial massage with the head of the therapeutic ultrasound device — Superficial massage with the head of the therapeutic ultrasound device will be applied to participants' back for 15 minutes, 3 times a week for 4 weeks in this group.
  Arms: Superficial massage with the head of the therapeutic ultrasound device

SUMMARY:
Menopause is defined as the permanent cessation of menstruation as a result of the loss of ovarian follicular function. This process involves some bothersome physical and psychological climacteric symptoms. The most common symptoms are vasomotor symptoms, psychological symptoms and sleep disturbances.

The aim of this study is to investigate the effects of CTM on postmenopausal symptoms, menopause-specific quality of life (MENQoL) and insomnia.

For this purpose, 58 postmenopausal women who meet the inclusion criteria and volunteer to participate in the study will be randomly assigned to one of the two research arms; CTM or sham control. The participants in the experimental group will receive CTM for 5-20 minutes, 3 times a week for 4 weeks, whereas the participant in the sham control group will receive superficial massage with the head of the therapeutic ultrasound device for 15 minutes at the same frequency for 4 weeks. In this study, primary outcome is menopausal symptom severity and will be assessed by the "Menopause Rating Scale". Secondary outcomes are hot flash frequency, hot flash score (frequency X severity), menopause-specific quality of life, emotional status and insomnia. These outcomes will be assessed by daily diaries and the questionnaires; "Menopause-Specific Quality of Life Scale", "Depression-Anxiety-Stress 21 Scale" and "Insomnia Severity Index". All outcome measurements will be evaluated at baseline and after the intervention period. Then, the results will be compared within groups and between two study groups.

DETAILED DESCRIPTION:
Menopause is defined as the permanent cessation of menstruation as a result of the loss of ovarian follicular function. It is part of the natural aging process and occurs by declining the estrogen secretion from the ovaries. This process involves some bothersome physical and psychological climacteric symptoms that negatively influence the women's well-being and quality of life. The most common symptoms are vasomotor symptoms (hot flashes, sweating, night sweats), psychological symptoms (anxiety, depression, stress) and insomnia. Although hormonal and non-hormonal pharmacological methods are widely used effective approaches to control these symptoms, they have some risks or adverse side effects. For this reason, women tend to alternative therapies and complementary medicine methods to improve climacteric symptoms and their quality of life.

Connective tissue manipulation (CTM) is a manual reflex therapy method which aims to restore the balance between the sympathetic and parasympathetic components of the autonomic nervous system. It is characterised by special type of manual stroke which is applied to the connective tissue. These stretching maneuvers are applied to areas called "reflex zones", and create local, segmental and general therapeutic effects in the body.

The aim of this study is to investigate the effects of CTM on postmenopausal symptoms, menopause-specific quality of life (MENQoL) and insomnia.

For this purpose, 58 postmenopausal women ages between 45 to 65 who meet the inclusion criteria and volunteer to participate in the study will be randomly assigned to one of the two research arms, CTM or sham control. The women in the experimental group will receive CTM for 5-20 minutes, 3 times a week for 4 weeks. On the other hand, the women in the sham control group will receive superficial massage with the head of the therapeutic ultrasound device for 15 minutes at the same frequency for 4 weeks. In this study, primary outcome is menopausal symptom severity and it will be evaluated by "Menopause Rating Scale". Secondary outcomes are hot flash frequency, hot flash score (frequency X severity), menopause-specific quality of life, emotional status and insomnia. These outcomes will be assessed by daily diaries and the questionnaires "Menopause-Specific Quality of Life Scale", "Depression-Anxiety-Stress 21 Scale" and "Insomnia Severity Index".

The diaries will be filled out for one week (7 days each); at the baseline and just after the completion of the study. All other outcome measurements will be performed before and immediately after the study is completed. The results will be compared within groups and between two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged between the 45 and 65 years,
* Being experienced at least 3 moderate or severe hot flashes, sweating or night sweats per day for at least 3 months,
* Being in the natural/spontaneous postmenopausal (amenorrhea for at least 12 months) period for less than 10 years,
* Having stable vital signs (heart rate, blood pressure),
* Volunteer to participate in the study,
* Have signed the informed consent form.

Exclusion Criteria

* Neurological diseases,
* Uncontrolled systemic and metabolic diseases (uncontrolled diabetes mellitus, hypertension, etc.)
* History of cancer,
* History of surgical menopause,
* Obesity (BMI > 35 kg/m²),
* Use of any hormonal or non-hormonal treatment for vasomotor or other menopausal symptoms in the past 6 months,
* Psychiatric and mental disorders that prevent the cooperation to the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Severity of menopausal symptoms | Change in the severity of menopausal symptoms from baseline to at the end of the 4th week.
  The severity of menopausal symptoms will be evaluated with the Menopause Rating Scale (MRS). MRS was developed to assess the severity of 11 symptoms associated with menopause. Each of the 11 symptoms may score between 0 (no symptoms) and 4 points (severe symptoms), depending on the perceived severity of the complaints. The total score of the MRS ranges between 0 (asymptomatic) and 44 (highest degree of complaints).

SECONDARY OUTCOMES:
Frequency of vasomotor symptoms | Change in the frequency of vasomotor symptoms from baseline to at the end of the 4th week.
  Frequency of hot flashes, sweating and night sweats will be assessed by daily diaries. Participants will record their hot flashes, sweating and night sweats during seven days at the baseline and just after the completion of the study.
Vasomotor symptom intensity | Change in the vasomotor symptom score from baseline to at the end of the 4th week.
  The vasomotor symptom intensity, which will be obtained by multiplying the frequency and severity (mild, moderate, severe) of hot flashes, sweating and night sweats assessed by daily diaries. Participants will record their hot flashes, sweating and night sweats during seven days at the baseline and just after the completion of the study.
Quality of life associated with menopause | Change in quality of life associated with menopause from baseline to at the end of the 4th week.
  Menopause-related quality of life will be assessed with the Menopause Specific Quality of Life Questionnaire (MENQOL). MENQOL was developed to determine how changes in the physical, psychological and social areas during the menopausal period affect the quality of life of women. The scale is an eight-point Likert-type scale and consists of 29 questions.
Level of psychological symptoms | Change in the level of psychological symptoms from baseline to at the end of the 4th week.
  The level of psychological symptoms will be evaluated with the Depression, Anxiety and Stress Scale-21 (DASS-21). DASS-21 is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
Severity of insomnia | Change in severity of insomnia from baseline to at the end of the 4th week.
  Severity of insomnia will be evaluated with the Insomnia Severity Index (ISI). ISI is a seven-item, five-point Likert-type questionnaire to assess the severity of sleep disturbance during the past two weeks. Total scores range from 0 to 28, with higher combined scores indicating worse insomnia severity.

OTHER OUTCOMES:
Intervention Satisfaction | Satisfaction with CTM and with placebo therapeutic ultrasound is compared at the end of the 4th week.
  Individual's satisfaction with CTM or placebo therapeutic ultrasound was assessed with the Visual Analog Scale (VAS). The "0" point at the left end of the 10 cm horizontal VAS was defined as "not at all satisfied", while the "10" point at the right end was defined as "very satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Serap Özgül, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gracia CR, Freeman EW. Onset of the Menopause Transition: The Earliest Signs and Symptoms. Obstet Gynecol Clin North Am. 2018 Dec;45(4):585-597. doi: 10.1016/j.ogc.2018.07.002. Epub 2018 Oct 25. PMID 30401544
- [Background] Roberts H, Hickey M. Managing the menopause: An update. Maturitas. 2016 Apr;86:53-8. doi: 10.1016/j.maturitas.2016.01.007. Epub 2016 Jan 22. PMID 26921929
- [Background] Santoro N, Epperson CN, Mathews SB. Menopausal Symptoms and Their Management. Endocrinol Metab Clin North Am. 2015 Sep;44(3):497-515. doi: 10.1016/j.ecl.2015.05.001. PMID 26316239
- [Background] Cobin RH, Goodman NF; AACE Reproductive Endocrinology Scientific Committee. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY POSITION STATEMENT ON MENOPAUSE-2017 UPDATE. Endocr Pract. 2017 Jul;23(7):869-880. doi: 10.4158/EP171828.PS. PMID 28703650
- [Background] Holey LA, Dixon J. Connective tissue manipulation: a review of theory and clinical evidence. J Bodyw Mov Ther. 2014 Jan;18(1):112-8. doi: 10.1016/j.jbmt.2013.08.003. Epub 2013 Sep 8. PMID 24411158
- [Background] Fu P, Gibson CJ, Mendes WB, Schembri M, Huang AJ. Anxiety, depressive symptoms, and cardiac autonomic function in perimenopausal and postmenopausal women with hot flashes: a brief report. Menopause. 2018 Dec;25(12):1470-1475. doi: 10.1097/GME.0000000000001153. PMID 29916944
- [Background] Guttuso T Jr, DiGrazio WJ, Reddy SY. Review of hot flash diaries. Maturitas. 2012 Mar;71(3):213-6. doi: 10.1016/j.maturitas.2011.12.003. Epub 2012 Jan 9. PMID 22230663
- [Background] Schneider HP, Heinemann LA, Rosemeier HP, Potthoff P, Behre HM. The Menopause Rating Scale (MRS): reliability of scores of menopausal complaints. Climacteric. 2000 Mar;3(1):59-64. doi: 10.3109/13697130009167600. PMID 11910611
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Derived] Albayrak G, Cagliyan Turk A, Ozgul S. Effects of connective tissue massage on physical and emotional symptoms, insomnia, and quality of life in postmenopausal women: A randomized, sham-controlled trial. Maturitas. 2025 Jan;191:108149. doi: 10.1016/j.maturitas.2024.108149. Epub 2024 Nov 7. PMID 39522476